CLINICAL TRIAL: NCT02970812
Title: Effects of Electrical Muscle Stimulation on Waist Circumference in Adults: A Randomized Controlled Trial
Brief Title: Effects of Electrical Muscle Stimulation on Waist Circumference in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003011
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical Muscle Stimulation (Experimental): Electrical Muscle Stimulation (EMS) program was consisted of warm-up, warm-down, contraction and relaxation. It was programed to be resemble to actual muscle action of voluntary exercise. To increase energy consumption as high intensity exercise, tripled the contraction duration. EMS group used Program 3 and regulated intensity though channel from 1 to 4.
  Interventions: Device: Electrical Muscle Stimulation
- Transcutaneous Electrical Nerve Stimulation (Placebo Comparator): Transcutaneous group used Transcutaneous Electrical Nerve Stimulation (TENS) which is the use of electric current produced to stimulate the sensory nerves to block pain signal. It is programed to applied currents regularly, once a second with a frequency of 1 Hz.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Electrical Muscle Stimulation — Participants were under EMS 5 times a week for 12 weeks. Pads were applied on participants' abdomen, rectus abdominis and external oblique abdominal muscle areas without any recent wound, infection, scar, and warts while lie on their back.
  Arms: Electrical Muscle Stimulation
Device: Transcutaneous Electrical Nerve Stimulation — Participants were under TENS 5 times a week for 12 weeks. Pads were applied on participants' abdomen, rectus abdominis and external oblique abdominal muscle areas without any recent wound, infection, scar, and warts while lie on their back.
  Arms: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
This randomized, placebo-controlled, double-blind, controlled study was designed to investigate the efficacy of electrical muscle simulation (EMS) for treatment of waist circumference (WC) reduction in abdominal obese adults.

60 patients with abdominal obese, man with WC > 90 cm and woman with WC > 80 cm, received EMS as experimental group (EG) or transcutaneous electrical nerve stimulation (TENS) as control group (CG) 5 times a week for 12 weeks.

DETAILED DESCRIPTION:
Background: This randomized, placebo-controlled, double-blind, controlled study was designed to investigate the efficacy of electrical muscle simulation (EMS) for treatment of waist circumference (WC) reduction in abdominal obese adults.

Methods: 60 patients with abdominal obese, man with WC > 90 cm and woman with WC > 80 cm, received EMS as experimental group (EG) or transcutaneous electrical nerve stimulation (TENS) as control group (CG) 5 times a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has abdominal obese seventy subjects between the age 18 and 65 years
* Abdominal obesity was defined as having a waist circumference (WC) >90 cm for men or WC >80 cm for women was defined based on the Asia-Pacific criteria of the International Diabetes Federation.

Exclusion Criteria:

* pregnant or breastfeeding, had taken any treatment for weight loss or any medication known to affect weight
* had a weight loss of 3% or more in the preceding 3 months, had undergone any major surgery during the 1 year prior to study commencement
* had any inserted metallic materials including a pacemaker.
* aspartate aminotransferase or alanine aminotransferase of 100 mg/dL or more
* serum creatinine of 1.5 mg/dL or more
* a history of coronary arterial disease or cerebrovascular disease, impairment of a major organ system, cancer, severe lung diseases, severe cerebral trauma, uncontrolled hypertension and psychiatric diseases including eating disorder, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrical Muscle Stimulation: EMS program was consisted of warm-up, warm-down, contraction and relaxation. It was programed to be resemble to actual muscle action of voluntary exercise. To increase energy consumption as high intensity exercise, tripled the contraction duration. EMS group used Program 3 and regulated intensity though channel from 1 to 4.
  EMS: Participants were under EMS 5 times a week for 12 weeks. Pads were applied on participants' abdomen, rectus abdominis and external oblique abdominal muscle areas without any recent wound, infection, scar, and warts while lie on their back.
- Electrical Nerve Stimulation: Transcutaneous group used Transcutaneous Electrical Nerve Stimulation (TENS) which is the use of electric current produced to stimulate the sensory nerves to block pain signal. It is programed to applied currents regularly, once a second with a frequency of 1 Hz.
  TENS: Participants were under TENS 5 times a week for 12 weeks. Pads were applied on participants' abdomen, rectus abdominis and external oblique abdominal muscle areas without any recent wound, infection, scar, and warts while lie on their back.
Period: Overall Study
Arm/Group | Electrical Muscle Stimulation | Electrical Nerve Stimulation
Started | 30 | 30
Completed | 22 | 28
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Muscle Stimulation | Electrical Nerve Stimulation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12.9) | 38.5 (10.6) | 39 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  South Korea | 30 | 30 | 60
Waist circumference [Mean (Standard Deviation); unit: cm] | 92.2 (11.6) | 92.3 (7.2) | 92.2 (9.6)
CT visceral fat [Mean (Standard Deviation); unit: cm^2] | 105.7 (66.3) | 91.0 (48.3) | 95.2 (58.1)

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference
Description: Waist circumference was measured by a tape
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Electrical Muscle Stimulation | Electrical Nerve Stimulation
Number analyzed (Participants) | 30 | 30
cm | 87.0 (12.4) | 89.4 (9.5)

ADVERSE EVENTS:
Time Frame: 3 months
Description: not-occurred
Arm/Group | Electrical Muscle Stimulation | Electrical Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No